CLINICAL TRIAL: NCT06929299
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of STSA-1301 Subcutaneous Injection in Healthy Subjects and Patients With Immune Thrombocytopenia (ITP)
Brief Title: A Phase Ib/II Clinical Trial of Multiple Doses of STSA-1301 Subcutaneous Injection in Healthy Subjects and Patients With Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu BioJeTay Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1301-02
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose of STSA-1301 subcutaneous injection or Placebo (First cohort) (Experimental)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- Median dose of STSA-1301 subcutaneous injection or Placebo (Second cohort) (Experimental)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- High dose of STSA-1301 subcutaneous injection or Placebo (Third cohort) (Experimental)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1301 subcutaneous injection — Subjects will receive the STSA-1301 on the dates specified in the protocol
Drug: Placebo — Subjects will receive the placebo on the dates specified in the protocol

SUMMARY:
A randomized, double-blind, placebo-controlled design was designed to evaluate the safety and tolerability, pharmacokinetic/pharmacodynamic profile, and immunogenicity of multiple administration of STSA-1301 subcutaneous injection in healthy subjects and patients with ITP, and to further explore the initial efficacy of STSA-1301 subcutaneous injection in patients with ITP

ELIGIBILITY:
Inclusion Criteria:

- (stage I):

1. 18 years ≤ age ≤ 50 years, male or female subjects;
2. Body mass index is 18 kg/m^2≤ BMI≤ 26kg/m^2;
3. Subjects (including the subject's partner) are willing to use effective contraception during the study period and have no plans to have children or to donate sperm or eggs from the time of signing the informed consent form until 3 months after the last dose;
4. Pre-randomization medical history had no effect on enrollment in the trial, and physical examination, laboratory test items, and all tests related to the trial were normal or the investigator determined that the abnormalities were not clinically significant;
5. Subjects are aware of the risks of the trial and voluntarily participate in this clinical trial and sign an informed consent form.

(stage 2):

1. Aged 18 to 75 years, inclusive, and of either gender.
2. Clinically diagnosed with persistent or chronic primary immune thrombocytopenia (ITP) with no known other causes of thrombocytopenia.
3. The ITP diagnosis of the subject is supported by a prior response to ITP treatment with a platelet count reaching ≥50×10^9/L.
4. One platelet test during the screening period and one during the baseline period (with an interval of at least 7 days), with an average platelet count <30×10^9/L and no single platelet count >35×10^9/L. No severe bleeding within 4 weeks prior to the screening visit.
5. Subjects who have previously failed at least one first-line standard ITP treatment (corticosteroids and/or intravenous immunoglobulin) (defined as inability to maintain efficacy or relapse), or are intolerant to first-line standard treatment.
6. The study allows the concurrent use of the following ITP treatment medications at a stable dose: oral corticosteroids, danazol, dapsone, oral immunosuppressants (azathioprine, methotrexate, cyclosporine A, mycophenolate mofetil), or TPO-RA (limited to oral small molecule non-peptide). A stable dose means that the treatment dose and frequency have been stable for at least 4 weeks prior to randomization and are not expected to change during the study.
7. The subject (including the subject's partner) is willing to use effective contraception from the time of signing the informed consent form until 3 months after the last dose of study drug, and has no plans for pregnancy or sperm/egg donation during this period.
8. The subject fully understands and is able to comply with the requirements of the study protocol and voluntarily signs the informed consent form.

Exclusion Criteria:

- (stage I)

1. Subject has a history of serious medical conditions (including, but not limited to, gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, pulmonary, immunologic, psychiatric, or cardiovascular disorders) or any disease or sequela known to be likely to interfere with the absorption, distribution, metabolism, or excretion of the test drug;
2. Subjects with an active infection or with a serious infection (resulting in hospitalization or requiring parenteral antibiotic therapy) within 6 weeks prior to the first dose; subjects with a combination of clinically significant active or chronic uncontrolled bacterial, viral, or fungal infections at screening;
3. Subjects have a history of immunodeficiency;
4. Subjects had a history of malignant tumors;
5. Subjects who are hypersensitive to the product or any of its ingredients; history of eczema, asthma or other allergic diseases;
6. Current active tuberculosis, including pulmonary and extrapulmonary tuberculosis; tuberculosis-related imaging changes in the lungs (e.g., cavities, infiltrative lesions) detected by chest X-ray; and a history of close contact with an active case of tuberculosis in the past 1 year.
7. Subject's total IgG at Screening/Baseline is less than the lower limit of normal. Subject has an absolute neutrophil count <1.5X10^9/L and/or an absolute lymphocyte count <1.0× 10^9/L;
8. Positive Hepatitis B Surface Antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb), Hepatitis C Virus Antibody (Anti-HCV), Syphilis Specific Antibody, and Positive HIV Antibody (Anti-HIV);
9. Those with clinically significant abnormalities on electrocardiogram (ECG) examination as judged by the clinical investigator (one repeat is permitted to determine eligibility);
10. The subject has any condition that interferes with blood collection (including difficulties in blood sample collection, etc.);
11. Consumption of more than 5 cups of coffee, tea, or cola (150mL each) per day in the 3 months prior to screening;
12. Smoked more than 5 cigarettes or equivalent amount of tobacco per day in the 3 months prior to screening;
13. Regular drinkers in the 6 months prior to screening, i.e., more than 2 units of alcohol per day (1 unit = 360mL of beer or 45mL of spirits at 40% alcohol or 150mL of wine) in the 6-month period; and abnormal breath test results for alcohol during the Screening Period or Baseline Period;
14. Subjects with a history of substance abuse within 1 year prior to screening; positive urine substance abuse screen at baseline;
15. Blood loss or blood donation >400mL within 3 months prior to screening or history of blood transfusion or any blood product use within 3 months prior to enrollment;
16. Participation as a subject in any drug or vaccine or medical device clinical trial within 3 months prior to screening;
17. Vaccinated or scheduled to be vaccinated within 4 weeks prior to screening up to 3 months after the end of dosing;
18. Taken medications that may affect immune function within 6 months prior to screening or received any monoclonal antibody or biologic therapy within 3 months prior to screening and prescription/over-the-counter medications, herbs, or other supplements within 14 days prior to screening;
19. Women who are pregnant or breastfeeding;
20. Subjects who, in the opinion of the investigator, have any factors that make participation in this trial inappropriate.

(stage 2)

1. Thrombocytopenia associated with other conditions such as lymphoma, chronic lymphocytic leukemia, viral infections, hepatitis, induced or alloimmune thrombocytopenia, thrombocytopenia associated with abnormal bone marrow development, or hematopoietic stem cell transplantation.
2. Abnormalities in any of the following laboratory tests at screening or at baseline: a. Total IgG level < 6 g/L. b. International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (APTT) > 1.5 x ULN. c. Alanine aminotransferase (ALT) ≥ 3× ULN or aspartate aminotransferase (AST) ≥ 3× ULN.
3. Clinical evidence of significantly unstable or poorly controlled acute or chronic disease other than ITP (e.g., cardiovascular, pulmonary, hematologic, gastrointestinal, endocrine, hepatic, renal, neurologic, infectious, poorly controlled diabetes mellitus) present at the time of screening, recent major surgical procedures, or any other medical condition that, in the opinion of the investigator, may affect the results of the study or the safety of the subject.
4. Prior comorbidities or treatments: a. Use of anticoagulants (e.g., vitamin K antagonists, direct oral anticoagulants) or any medication with antiplatelet effects within 4 weeks prior to randomization. b. Any blood transfusion within 4 weeks prior to randomization. c. Received Ig (IV, SC, or intramyocardial routes) or plasma exchange (PLEX) or anti-D immunoglobulin therapy within 4 weeks prior to randomization. d. Use of recombinant human thrombopoietin or Romiplostim within 6 months prior to randomization. e. Use of rituximab or other anti-CD20 agents other than rituximab within 6 months prior to randomization. f. Splenectomy within 3 months prior to randomization. g. Live/attenuated vaccine within 8 weeks prior to randomization. h. Vaccination within 8 weeks prior to randomization. i. Vaccination within 8 weeks prior to randomization. j. Vaccination within 8 weeks prior to screening. k. Receipt of any inactivated, subunit, polysaccharide, or conjugate vaccine at any time prior to screening is not considered an exclusion criterion. h. Use of other complementary therapies that have been evaluated by the investigator at as potentially interfering with the subject's efficacy assessment and safety, including but not limited to: herbal medicines, herbal remedies, or manipulations (e.g., acupuncture) within the greater of 4 weeks or 5 half-lives prior to randomization.
5. Prior history of malignancy, except for cured carcinoma in situ.
6. Any thrombotic or embolic event within 12 months prior to randomization, or history of any major thrombotic or embolic event within 5 years (e.g., myocardial infarction, stroke, deep vein thrombosis, or pulmonary embolism).
7. History of coagulation disorders or hereditary thrombocytopenia or family history of thrombocytopenia.
8. Presence of active, clinically significant organ or internal mucosal bleeding requiring urgent treatment or therapeutic manipulation (e.g., intracranial hemorrhage, pulmonary hemorrhage, hemorrhage persistently requiring transfusion of concentrated red blood cells) within 6 months prior to screening.
9. In the judgment of the investigator, it is predicted that there may be a higher risk of clinically significant organ or internal mucosal hemorrhage requiring urgent treatment or therapeutic manipulation during the study period (e.g., intracranial hemorrhage, pulmonary hemorrhage, hemorrhage that consistently requires transfusion of concentrated red blood cells).
10. Presence of clinically significant active or chronic bacterial, viral, or fungal infections at screening or at baseline; or acute or chronic infectious diseases requiring systemic therapy with antibiotics, antivirals, antiparasitics, or antifungals within 4 weeks prior to randomization.
11. Hepatitis B surface antigen (HBsAg) positive at screening, or hepatitis B core antibody (HBcAb) positive+ Hepatitis B virus deoxyribonucleic acid (HBV-DNA) positive, or hepatitis C virus (HCV) antibody positive+ Hepatitis C virus ribonucleic acid (HCV-RNA) positive, or human immunodeficiency virus (HIV) antibody or syphilis antibody positive.
12. Currently has active tuberculosis, including pulmonary and extrapulmonary tuberculosis; chest X-ray reveals tuberculosis-related imaging changes in the lungs (e.g., cavities, infiltrative lesions).
13. Hypersensitivity reactions to the study drug are known to exist.
14. Participated in a clinical study of another FcRn inhibitor in the previous 6 months and received at least 1 administration.
15. Have used the investigational drug within 3 months or 5 half-lives (whichever is longer) prior to randomization.
16. Being pregnant or breastfeeding at screening or at baseline or having plans to become pregnant during the study.
17. Presence of an autoimmune disease other than ITP at screening or at baseline.
18. Other conditions that, in the judgment of the investigator, make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To Evaluate any adverse event that occurs in the subject after administration of the drug | 78 Days

SECONDARY OUTCOMES:
Pharmacodynamic (PD) indicators: Serum total IgG | 78 days
Proportion of subjects achieving a platelet count ≥30× 10^9/L at least 2 times within 11 weeks of the first administration of the drug | 78 days
Proportion of subjects achieving a response (R) within 11 weeks of first dosing | 78 days
Proportion of subjects achieving a complete response (CR) within 11 weeks of initial dosing | 78 days
Proportion of subjects achieving a platelet count ≥50× 10^9/L at least 2 times within 11 weeks of the first administration of the drug | 78 days
Onset time from first dose to first achieved platelet count ≥30× 10^9/L, 50× 10^9/L, or 100× 10^9/L | 78 days
Change from Baseline in Subject WHO Bleeding Score at 11 Weeks After Initial Dosing | 78 days
Immunogenicity indicators:Incidence of positive anti-drug antibodies (ADA) | 78 days
Cytokines: TNF-α, IL-6 | 78 days
Blood concentration and PK parameters :Cmax | 78 days
Blood concentration and PK parameters : Cmin | 78 days
Blood concentration and PK parameters : AUC0-t | 78 days
Blood concentration and PK parameters: AUClast | 78 days
Blood concentration and PK parameters: AUC0-∞ | 78 days
Blood concentration and PK parameters: Tmax | 78 days
Blood concentration and PK parameters: t1/2 | 78 days
Blood concentration and PK parameters: kel | 78 days
Blood concentration and PK parameters: CL/F | 78 days
Blood concentration and PK parameters: VZ/F | 78 days
Blood concentration and PK parameters: MRTlast | 78 days
Blood concentration and PK parameters: Rac | 78 days

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D., Principal Investigator — Hospital of Hematology, Chinese Academy of Medical Sciences; Yi Fang, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (7):
- China (7):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality